CLINICAL TRIAL: NCT01291147
Title: Local Anaesthetic Infusion For Laparoscopic Hysterectomy: A Randomised Controlled Trial
Brief Title: Local Anaesthetic Infusion For Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ashford and St. Peter's Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010JTW01
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Postoperative Pain
Keywords: pain; anaesthetic
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levobupivicaine (Active Comparator)
  Interventions: Drug: Levobupivicaine
- 0.9% Saline (Placebo Comparator)
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: Levobupivicaine — levobupivicaine 0.5% continous infusion for 48 hours
  Arms: Levobupivicaine
Drug: 0.9% Saline — 0.9% saline continous infusion for 48 hours
  Arms: 0.9% Saline

SUMMARY:
More hysterectomies are performed laparoscopically either as a total laparoscopic hysterectomy or as a laparoscopically assisted vaginal hysterectomy. The advantages of laparoscopic surgery include quicker hospital discharge, a shorter convalescence and cost effectiveness when compared to open procedures. Laparoscopic hysterectomies (both total and vaginally assisted) can lead to discomfort which may lead to a delay in discharge from hospital. Continuous infusions of local anaesthetic agents given post operatively to the site of operation have the been subject of trials for several operative procedures. To date however there have not been any properly controlled studies evaluating whether there are benefits of giving a local anaesthetic infusion for 48 hours into the pelvis following a total or vaginally assisted laparoscopic hysterectomy. The investigators therefore propose to investigate whether giving a local anaesthetic infusion in this fashion decreases the amount of rescue and patient controlled analgesia needed, and length of hospital stay. In order to do this the investigators wish to conduct a randomised placebo controlled double blind trial.

ELIGIBILITY:
Inclusion Criteria:

All women undergoing a total laparoscopic or laparoscopically assisted vaginal hysterectomy

Exclusion Criteria:

Women undergoing surgery for cancer, or are known to be allergic to local anaesthetic agents.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
• Need for 'rescue' analgesia | 48 hours

SECONDARY OUTCOMES:
• Pain intensity | 48 hours
Side effects from rescue analgesia | 48 hours
Amount of patient controlled analgesia needed | 48 hours
Hospital length of stay | 48 hours
Patient satisfaction with pain relief | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy T Wright, MD FRCOG, Principal Investigator — Ashford and St Peter's Hospitals NHS Foundation Trust
Locations (1):
- Ashford and St Peter's Hospitals NHS Foundation Trust, Chertsey, Surrey, United Kingdom

REFERENCES:
- [Derived] Andrews V, Wright JT, Zakaria F, Banerjee S, Ballard K. Continuous infusion of local anaesthetic following laparoscopic hysterectomy--a randomised controlled trial. BJOG. 2014 May;121(6):754-60; discussion 761. doi: 10.1111/1471-0528.12610. Epub 2014 Feb 19. PMID 24548730